CLINICAL TRIAL: NCT03481777
Title: Remote Ischemic Conditioning in Patients With Acute Stroke: a Multicenter Randomized, Patient-assessor Blinded, Sham-controlled Study
Brief Title: Remote Ischemic Conditioning in Patients With Acute Stroke (RESIST)
Acronym: RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grethe Andersen (Other)
Collaborators: Danish National Research Foundation (Other); Central Denmark Region (Other)
Responsible Party: Sponsor-Investigator, Grethe Andersen, Professor, DMSc, Senior Consultant, MD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017114177
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute; Ischemic Stroke; Hemorrhagic Stroke; Intracerebral Hemorrhage; Cerebrovascular Disorders; Central Nervous System Diseases
Keywords: Remote Ischemic Conditioning; Neuroprotection
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebral Hemorrhage; Cerebrovascular Disorders; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, patient-assessor blinded, sham-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant. Outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (Active Comparator): Remote ischemic conditioning (RIC) is applied in the hyperacute prehospital phase using an automated RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be 200 mmHg; but if initial systolic blood pressure is above 175 mmHg, the cuff is automatically inflated to 35 mmHg above the systolic blood pressure.
  * Initial remote ischemic conditioning: prehospital phase, all included patients
  * Remote ischemic conditioning at +6 hours: In-hospital, only patients with AIS and ICH, all centres
  * Remote Ischemic Postconditioning (twice daily for 7 days): In-hospital/rehabilitation, Only patients with AIS and ICH and only at Aarhus University Hospital
  Usual care with or without acute reperfusion therapy
  Interventions: Device: Remote Ischemic Conditioning
- Sham - Remote Ischemic Conditioning (Sham Comparator): Sham remote ischemic conditioning (Sham-RIC) is applied in the hyperacute prehospital phase using an automated Sham-RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be always be 20 mmHg.
  * Initial Sham remote ischemic conditioning: prehospital phase, all included patients
  * Sham Remote ischemic conditioning at +6 hours: In-hospital, only patients with AIS and ICH, all centres
  * Sham Remote Ischemic Postconditioning (twice daily for 7 days): In-hospital/rehabilitation, Only patients with AIS and ICH and only at Aarhus University Hospital
  Usual care with or without acute reperfusion therapy.
  Interventions: Device: Sham Remote Ischemic Conditioning

INTERVENTIONS:
Device: Remote Ischemic Conditioning — RIC is commonly achieved by inflation of a blood pressure cuff to induce 5-minute cycles of limb ischemia alternating with 5 minutes of reperfusion.
  Arms: Remote Ischemic Conditioning
Device: Sham Remote Ischemic Conditioning — Sham Comparator (Sham-RIC)
  Arms: Sham - Remote Ischemic Conditioning

SUMMARY:
Our primary aim is to investigate whether remote ischemic conditioning (RIC) as an adjunctive treatment can improve long-term recovery in acute stroke patients as an adjunct to standard treatment.

DETAILED DESCRIPTION:
Stroke is the second-leading cause of death worldwide and a leading cause of serious, long-term disability. The most common type is acute ischemic stroke (AIS) which occurs in 85% of cases. Acute cerebral thromboembolism leads to an area of permanent damage (infarct core) in the most severely hypoperfused area and a surrounding area of impaired, yet salvageable tissue known as the "ischemic penumbra".

Intravenous alteplase (IV tPA) and endovascular treatment (EVT) are approved acute reperfusion treatments of AIS to be started within the first 4½-6 hours (in some up to 24 hours) and as soon as possible after symptom onset to prevent the evolution of the infarct core. However, reperfusion itself may paradoxically result in tissue damage (reperfusion injury) and may contribute to infarct growth. Infarct progression can continue for days following a stroke, and failure of the collateral flow is a critical factor determining infarct growth.

On the other hand, in intracerebral hemorrhage (ICH) the culprit is an eruption of blood into the brain parenchyma causing tissue destruction with a massive effect on adjacent brain tissues. Hematoma expansion as well as inflammatory pathways that are activated lead to further tissue damage, edema, and penumbral hypoperfusion. The prognosis after ICH is poor with a one-month mortality of 40%.

Novel therapeutics and neuroprotective strategies that can be started ultra-early after symptom onset are urgently needed to reduce disability in both AIS and ICH.

Ischemic conditioning is one of the most potent activators of endogenous protection against ischemia-reperfusion injury. Remote Ischemic Conditioning (RIC) can be applied as repeated short-lasting ischemia in a distant tissue that results in protection against subsequent long-lasting ischemic injury in the target organ. This protection can be applied prior to or during a prolonged ischemic event as remote ischemic pre-conditioning (RIPreC) and per-conditioning (RIPerC), respectively, or immediate after reperfusion as remote ischemic post-conditioning (RIPostC). RIC is commonly achieved by inflation of a blood pressure cuff to induce 5-minute cycles of limb ischemia alternating with 5 minutes of reperfusion.

Preclinical studies show that RIC induces a promising infarct reduction in an experimental stroke model. Results from a recent proof-of-concept study at our institution indicate that RIPerC applied during ambulance transportation as an adjunctive to in-hospital IV tPA increases brain tissue survival after one month. Furthermore, RIPerC patients had less severe neurological symptoms at admission and tended to have decreased perfusion deficits.

To-date, no serious adverse events have been documented in RIC.

RIC is a non-pharmacologic and non-invasive treatment without noticeable discomfort that has first-aid potential worldwide. However, whether combined remote ischemic per- and postconditioning can improve long-term recovery in AIS and ICH has never been investigated in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (≥ 18 years)
* Prehospital putative stroke (Prehospital Stroke Score, PreSS >= 1)
* Onset of stroke symptoms < 4 hours before RIC/Sham-RIC
* Independent in daily living before symptom onset (mRS ≤ 2)

Exclusion Criteria:

* Intracranial aneurisms, intracranial arteriovenous malformation, cerebral neoplasm or abscess
* Pregnancy
* Severe peripheral arterial disease in the upper extremities
* Concomitant acute life-threatening medical or surgical condition
* Arteriovenous fistula in the arm selected for RIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, MD, DMSc, Principal Investigator — Aarhus University Hospital, Department of Neurology
Locations (4):
- Denmark (4):
  - Department of Neurology Aarhus University Hospital, Aarhus, Danmark
  - Aalborg University Hospital, Aalborg, DK
  - Odense University Hospital, Odense, DK
  - Department of Neurology Regional Hospital West Jutland, Holstebro

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following arcticle publication
Access Criteria: Proprosals should be directed to rolfblau@rm.dk. To gain access data requestors will need to sign a data processing agreement.

REFERENCES:
- [Background] Hess DC, Blauenfeldt RA, Andersen G, Hougaard KD, Hoda MN, Ding Y, Ji X. Remote ischaemic conditioning-a new paradigm of self-protection in the brain. Nat Rev Neurol. 2015 Dec;11(12):698-710. doi: 10.1038/nrneurol.2015.223. Epub 2015 Nov 20. PMID 26585977
- [Background] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Background] Blauenfeldt RA, Hjort N, Gude MF, Behrndtz AB, Fisher M, Valentin JB, Kirkegaard H, Johnsen SP, Hess DC, Andersen G. A multicentre, randomised, sham-controlled trial on REmote iSchemic conditioning In patients with acute STroke (RESIST) - Rationale and study design. Eur Stroke J. 2020 Mar;5(1):94-101. doi: 10.1177/2396987319884408. Epub 2019 Oct 25. PMID 32232175
- [Result] Blauenfeldt RA, Hjort N, Valentin JB, Homburg AM, Modrau B, Sandal BF, Gude MF, Hougaard KD, Damgaard D, Poulsen M, Diedrichsen T, Schmitz ML, von Weitzel-Mudersbach P, Christensen AA, Figlewski K, Grove EL, Hreietharsdottir MK, Lassesen HM, Wittrock D, Mikkelsen S, Vaeggemose U, Juelsgaard P, Kirkegaard H, Rostgaard-Knudsen M, Degn N, Vestergaard SB, Damsbo AG, Iversen AB, Mortensen JK, Petersson J, Christensen T, Behrndtz AB, Botker HE, Gaist D, Fisher M, Hess DC, Johnsen SP, Simonsen CZ, Andersen G. Remote Ischemic Conditioning for Acute Stroke: The RESIST Randomized Clinical Trial. JAMA. 2023 Oct 3;330(13):1236-1246. doi: 10.1001/jama.2023.16893. PMID 37787796
- [Result] Blauenfeldt RA, Simonsen CZ, Valentin JB, Johnsen SP, Hjort N, Andersen G. Outcomes Following Adherence to a Randomized Stroke Trial Protocol. JAMA Netw Open. 2024 Jan 2;7(1):e2349730. doi: 10.1001/jamanetworkopen.2023.49730. PMID 38165678
- [Result] Blauenfeldt RA, Mortensen JK, Hjort N, Valentin JB, Homburg AM, Modrau B, Sandal BF, Gude MF, Berhndtz AB, Johnsen SP, Hess DC, Simonsen CZ, Andersen G. Effect of Remote Ischemic Conditioning in Ischemic Stroke Subtypes: A Post Hoc Subgroup Analysis From the RESIST Trial. Stroke. 2024 Apr;55(4):874-879. doi: 10.1161/STROKEAHA.123.046144. Epub 2024 Feb 1. PMID 38299363
- [Derived] Ganesh A, Gaist D, Modrau B, Gude MF, Behrndtz AB, Andersen G, Simonsen CZ, Blauenfeldt RA. Pre-hospital treatment duration and efficacy of remote ischaemic conditioning in the RESIST randomised-controlled trial. Eur Stroke J. 2026 Jan 1;11(1):aakaf015. doi: 10.1093/esj/aakaf015. PMID 41614496
- [Derived] Blauenfeldt RA, Hess DC, Gaist D, Modrau B, Valentin JB, Johnsen SP, Hjort N, Behrndtz AB, Gude MF, Zhao W, Jensen J, Andersen G, Simonsen CZ. The Effect of Remote Ischemic Conditioning in Patients Treated with Endovascular Therapy: A RESIST Trial Post Hoc Study. Transl Stroke Res. 2025 Dec;16(6):2173-2184. doi: 10.1007/s12975-025-01379-5. Epub 2025 Sep 6. PMID 40913213
- [Derived] Blauenfeldt RA, Waller J, Drasbek KR, Bech JN, Hvas AM, Larsen JB, Andersen MN, Nielsen MC, Kjolhede M, Kjeldsen M, Gude MF, Khan MB, Baban B, Andersen G, Hess DC. Effect of Remote Ischemic Conditioning on the Form and Function of Red Blood Cells in Patients With Acute Ischemic Stroke. Stroke. 2025 Mar;56(3):603-612. doi: 10.1161/STROKEAHA.124.048976. Epub 2025 Jan 30. PMID 39882626

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The RESIST trial is a prehospital stroke trial. Patients are randomzied to remote ischemic conditioning or sham in the ambualnce before their final diagnosis. Patients who have a stroke (ischemic stroke or intracerebral hemorrhage, n= 902) are the target population and treated further according to randomization and outcome assessed as 3 months modified Rankin Scale . Patients with a non stroke diagnosis (n=531) are not treated further and not followed beyond hospital discharge.
Groups:
- Remote Ischemic Condtioning (RIC); Sham Remote Ischemic Conditioning: Patients with a prehospital stroke suspicion were randomized and treated with either RIC or sham RIC in the ambulance and continued at the stroke center. Patients with a in-hospital diagnosis of acute ischemic stroke or intracerebral hemorrhage were the target group and study population for the primary endpoint (modified Intention to Treat)
Period: Overall Study
Arm/Group | Remote Ischemic Condtioning (RIC) | Sham Remote Ischemic Conditioning
Started | 749 | 751
Completed | 436 (1500 (with suspected stroke) were randomized in the ambulance and of these 902 had a in-hospital target diagnosis of acute stroke) | 466
Not Completed | 313 | 285
Not completed — Withdrawal by Subject | 36 | 31
Not completed — Non stroke = non target population | 277 | 254

BASELINE CHARACTERISTICS:
Groups:
- Remote Ischemic Conditioning: Remote Ischemic Conditioning (Active)
- Sham: Remote Ischemic Conditioning (Sham)
- Total: Total of all reporting groups
Arm/Group | Remote Ischemic Conditioning | Sham | Total
Number analyzed (Participants) | 436 | 466 | 902
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [62 to 79] | 73 [62 to 80] | 73 [62 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 170 | 335
  Male | 271 | 296 | 567
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 436 | 466 | 902
National Institutes of Health Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: points on NIHSS] — Range 0-42, higher scores indicating more severe neurological symptoms
  points on NIHSS | 5 [2 to 11] | 5 [2 to 10] | 5 [2 to 10]
Diagnosis [Count of Participants; unit: Participants]
  Acute ischemic stroke | 349 | 388 | 737
  Intracerebral hemorrhage | 87 | 78 | 165

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale at 3 Months in Acute Stroke (AIS and ICH)
Description: Clinical outcome (modified Rankin Scale) at 3 months in acute stroke patients (target diagnosis) (generalized ordinal logistic regression). The assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death)
  If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  * If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  * If disagreement occurs between one face-to-face assessment and one telephone assessment
    * the face-to-face will be considered the final assessment
  * If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Remote Ischemic Conditioning (RIC): Patients with acute ischemic stroke or intracerbreral hemorrhage treated with Remote Ischemic Conditioning
- Sham: Patients with acute ischemic stroke or intracerbreral hemorrhage treated with Sham
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 436 | 466
units on a scale | 2 [1 to 3] | 1 [1 to 3]

2. Secondary Outcome: Difference Neurological Impairment During the First 24 Hours
Description: Neurological deficits are documented using Prehospital Stroke Score (PreSS). Prehospital Stroke Score is assessed in the the ambulance and at 24-hour or at discharge (if discharge occurs before 24 hours). The PreSS score consists of the Cincinnati Prehospital Stroke Scale (CPSS) with an additional opportunity to report other neurological symptoms (e.g. ataxia, sensory disturbances and visual field loss), and PASS (Prehospital Acute Stroke Severity Scale). The PreSS score range from 0-6, with 6 representing the most severe neurological deficits.
Time Frame: 24 hours
Population: 24-hour difference in prehospital stroke score
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Remote Ischemic Conditioning: Remote ischemic conditioning (RIC) is applied in the hyperacute prehospital phase using an automated RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be 200 mmHg; but if initial systolic blood pressure is above 175 mmHg, the cuff is automatically inflated to 35 mmHg above the systolic blood pressure.
  * Initial remote ischemic conditioning: prehospital phase, all included patients
  * Remote ischemic conditioning at +6 hours: In-hospital, only patients with AIS and ICH, all centres
  * Remote Ischemic Postconditioning (twice daily for 7 days): In-hospital/rehabilitation, Only patients with AIS and ICH and only at Aarhus University Hospital
  Usual care with or without acute reperfusion therapy
  Remote Ischemic Conditioning: RIC is commonly achieved by inflation of a blood pressure cuff to induce 5-minute cycles of limb ischemia alternating with 5 minutes of reperfusion.
- Sham - Remote Ischemic Conditioning: Sham remote ischemic conditioning (Sham-RIC) is applied in the hyperacute prehospital phase using an automated Sham-RIC device.
  Treatment characteristics: Five cycles (50 minutes), each consisting of five minutes of cuff inflation followed by five minutes with a deflated cuff. The cuff pressure will be always be 20 mmHg.
  * Initial Sham remote ischemic conditioning: prehospital phase, all included patients
  * Sham Remote ischemic conditioning at +6 hours: In-hospital, only patients with AIS and ICH, all centres
  * Sham Remote Ischemic Postconditioning (twice daily for 7 days): In-hospital/rehabilitation, Only patients with AIS and ICH and only at Aarhus University Hospital
  Usual care with or without acute reperfusion therapy.
  Sham Remote Ischemic Conditioning: Sham Comparator (Sham-RIC)
Arm/Group | Remote Ischemic Conditioning | Sham - Remote Ischemic Conditioning
Number analyzed (Participants) | 436 | 466
units on a scale | -1 [-2 to 0] | -2 [-2 to 0]

3. Secondary Outcome: Clinical Outcome (Modified Rankin Scale (mRS) at 3 Months in Acute Ischemic Stroke
Description: Clinical outcome (modified Rankin Scale) at 3 months in acute stroke patients (target diagnosis) (generalized ordinal logistic regression). TThe assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death) If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  If disagreement occurs between one face-to-face assessment and one telephone assessment the face-to-face will be considered the final assessment If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Population: Acute ischemic stroke patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Remote Ischemic Conditioning (RIC): Remote Ischemic Conditioning
- Sham: Sham
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 349 | 388
units on a scale | 1 [1 to 2] | 1 [0 to 3]

4. Secondary Outcome: Clinical Outcome (Modified Rankin Scale (mRS) at 3 Months in Acute Ischemic Stroke Receiving Reperfusion Therapy
Description: Clinical outcome (modified Rankin Scale) at 3 months inacute ischemic stroke receiving reperfusion therapy (generalized ordinal logistic regression). The assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death) If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  If disagreement occurs between one face-to-face assessment and one telephone assessment the face-to-face will be considered the final assessment If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Population: Patients with acute ischemic stroke who were treated with reperfusion therapies (intravenous thrombolysis and/or trombectomy)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 247 | 274
units on a scale | 1 [1 to 3] | 1 [1 to 3]

5. Secondary Outcome: Clinical Outcome (Modified Rankin Scale (mRS) at 3 Months in Patients With Intracerebral Hemorrhage (ICH)
Description: Clinical outcome (modified Rankin Scale) at 3 months in patients with intracerebral hemorrhage (ICH) (generalized ordinal logistic regression).
  The assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death) If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  If disagreement occurs between one face-to-face assessment and one telephone assessment the face-to-face will be considered the final assessment If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Population: Patients diagnosed with intracerebral hemorrhage
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 87 | 78
units on a scale | 3 [2 to 5] | 3 [2 to 5]

6. Secondary Outcome: Difference in Proportion of Patients With Complete Remission of Symptoms Within 24 Hours (TIA; Both With and Without DWI)
Description: Difference in proportion of patients with complete remission of symptoms within 24 hours (TIA; both with and without DWI) Diagnosis of TIA is documented in the electronic case report form
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 515 | 536
Participants | 96 | 90

7. Secondary Outcome: Major Adverse Cardiac and Cerebral Events (MACCE)
Description: MACCE is defined as: Cardiovascular events (cardiovascular death, myocardial infarction, acute ischemic or hemorrhagic stroke)
  Cardiovascular death: Death from known cardiovascular cause or sudden death from unknown cause (no identified cause of death in medical history and/or autopsy)
  Acute myocardial infarction: Admission with a discharge diagnosis of ST-elevation myocardial infarction (STEMI) and non-ST elevation myocardial infarction (NSTEMI) and unstable angina pectoris (UAP)
  Stroke: Admission with a discharge diagnosis of acute ischemic or hemorrhagic stroke. Evaluation is performed using the Danish National Patient Register (LPR) and the DSR at two time points (6 and 15 months after the inclusion of the last patient).
  Diagnosis of AIS/TIA, ICH and MI (STEMI, NSTEMI, and UAP) are made according to national clinical practice guidelines.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 436 | 466
Participants | 57 | 62

8. Secondary Outcome: Early Neurological Improvement in Acute Ischemic Stroke Patients (AIS)
Description: Reduction in National Institute of Health Stroke Scale (NIHSS) ≥ 4 (baseline versus 24-Hour NIHSS). NIHSS range from 0 to 42, with higher scores representing worse neurological function.
Time Frame: 24 hours
Population: Target population with acute stroke
Measure: Count of Participants; unit: Participants
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
Number analyzed (Participants) | 425 | 451
Participants | 108 | 131

9. Secondary Outcome: Early Neurological Improvement in Patients With Intracerebral Hemorrhage (ICH)
Description: as for outcome 8
Time Frame: 24 hours
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Quality of Life Measures at 3 Months in AIS and ICH Patients
Description: Quality of life (WHO-5 Well-Being Index) measures in AIS and ICH patients at 3 months
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2026-05

11. Secondary Outcome: Bed-day Use in AIS and ICH Patients
Description: Bed-day use, measured at 3 months, in AIS and ICH patients
Time Frame: 3 months
Reporting Status: Not Posted

12. Secondary Outcome: Three-month and One-year Mortality
Description: All-cause mortality is assessed and subdivided into cardiovascular mortality versus non-cardiovascular mortality
Time Frame: 3 and 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Clinical Outcome [Modified Rankin Scale (mRS) at 3 Months in Ischemic Stroke Patients and the Extended Remote Ischemic Postconditioning Protocol (Substudy at Aarhus University Hospital]
Description: Clinical outcome [modified Rankin Scale (mRS) at 3 months in ischemic stroke patients and the extended remote ischemic postconditioning protocol Ordinal logistic regression analysis will be performed.The assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death) If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  If disagreement occurs between one face-to-face assessment and one telephone assessment the face-to-face will be considered the final assessment If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2026-12

14. Other Pre Specified Outcome: Clinical Outcome (Modified Rankin Scale (mRS) at 3 Months in Intracerebral Hemorrhage Patients and the Extended Remote Ischemic Postconditioning Protocol (Substudy at Aarhus University Hospital)
Description: Clinical outcome (modified Rankin Scale (mRS) at 3 months in intracerebral hemorrhage patients and the extended remote ischemic postconditioning protocol The assessment will performed by two independent telephone or face-to-face assessors.
  the mRS range from 0 to 6, with higher scores representing worse outcome (mRS 0, no symptoms; mRS 6, death) If disagreement occurs the patient will be contacted by a third assessor (face-to-face or telephone) who is blinded to the intervention who will assess the level of dependency.
  If disagreement occurs between two telephone assessments - a third, and final, telephone or face-to-face assessment will be made.
  If disagreement occurs between one face-to-face assessment and one telephone assessment the face-to-face will be considered the final assessment If disagreement occurs between two face-to-face assessments - a third, and final, telephone or face-to-face assessment will be made.
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2026-12

15. Other Pre Specified Outcome: Endovascular Treatment(EVT) -Eligibility (MRI Assessed) in RIC Treated AIS Patients With Large Vessel (Substudy at Aarhus University Hospital)
Description: Proportion of RIC treated AIS patients with large vessel occlusion (LVO) eligible to EVT treatment compared to standard treatment, adjusted for prehospital stroke severity (PreSS) and symptom duration
  * Severe Stroke (NIHSS ≥ 10)
  * Groin puncture feasible within 6 hours from stroke onset
  * MRI-time-of-flight (TOF) documented internal carotid artery (ICA), Intracranial ICA (ICA-T) and first and second stem of the middle cerebral artery (M1 and M2, respectively)
  * No contraindications to MRI (pacemaker, vomiting, respiratory insufficiency, obesity)
  * MRI-Diffusion weighted imaging (DWI) lesion volume ≤ 70 mL
Time Frame: 6 hours
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Infarct Growth in AIS Patients (Substudy at Aarhus University Hospital)
Description: 24-hour infarct growth on DWI-MRI (Difference in lesion volume between acute and 24-hour DWI-MRI) (Substudy at Aarhus University Hospital)
Time Frame: 24 hour
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Difference in Acute (24-hour) Hematoma Expansion in Patients With ICH (Substudy at Aarhus University Hospital)
Description: 24-hour hematoma growth (Difference in hematoma volume between acute and 24-hour CT/MRI) (Substudy at Aarhus University Hospital)
Time Frame: 24 hour
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Difference in 7 Days Hematoma Volume in Patients With ICH (Substudy at Aarhus University Hospital)
Description: 7-day hematoma reduction (Difference in hematoma volume between acute and 7-day (day 5 to 9) CT ) (Substudy at Aarhus University Hospital)
Time Frame: 7 days
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Ektacytometry and Analytical Flow Cytometry for eryNOS3 Phosphorylation
Description: Ektacytometry for Erythrocytic Deformability and Analytical Flow Cytometry (FC) for eryNOS3 phosphorylation (pNOS3Ser1177) and s-nitrosylation (-SNO) in RBC
Time Frame: 12 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: MicroRNA and Extracellular Vesicle Profile of RIC-induced Neuroprotection
Description: MicroRNA and extracellular vesicle characterization of a possible RIC treatment profile (substudy at Aarhus University Hospital)
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

21. Other Pre Specified Outcome: Prehospital microRNA and Extracellular Vesicles (Substudy at Aarhus University Hospital)
Description: Diagnostic abilities of a prehospital microRNA and extracellular vesicles blood samples profile combined with prehospital stroke severity on the differentiation of hemorrhagic from ischemic stroke and to grade ischemic stroke severity
Time Frame: 12 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Prehospital Glial Fibrillary Acidic Protein (Substudy at Aarhus University Hospital)
Description: Predictive abilities of Glial Fibrillary Acidic Protein (GFAP) in prehospital obtained blood samples combined with prehospital stroke severity to differentiate hemorrhagic from ischemic stroke and to grade ischemic stroke severity
Time Frame: 12 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Coagulation Profile of Putative Stroke Patients in Prehospital Obtained Blood Samples
Description: Functional and immunologic plasma assays will be employed to analyze proteins and pathways in coagulation and fibrinolysis (substudy at Aarhus University Hospital)
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: 90 days
Description: Adverse events and adverse device events are defined according to ISO 14155:2011 and European Commission guideline on medical devices (MEDDEV 2.7/3 revision 3).
Arm/Group | Remote Ischemic Conditioning (RIC) | Sham
All-Cause Mortality (participants affected / at risk) | 41/713 | 47/720
Serious Adverse Events (participants affected / at risk) | 335/713 | 325/720
Other Adverse Events (participants affected / at risk) | 54/713 | 11/720
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Ischemic Conditioning (RIC) (N=713) | Sham (N=720)
SAE (Cardiac disorders) | 335 (335) | 325 (325) — All cause mortality
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Ischemic Conditioning (RIC) (N=713) | Sham (N=720)
Upper extremity pain during treatment and/or skin petechia (Musculoskeletal and connective tissue disorders) | 54 (54) | 11 (11) — Upper extremity pain during treatment and/or skin petechia for ALL randomized (Target diagnosis, non-target diagnosis and post-randomization exlcuded patients)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03481777/Prot_SAP_000.pdf